CLINICAL TRIAL: NCT05260242
Title: Delivering Empowering Conversations About Obstetric Regional Anesthesia for Underserved Minorities
Acronym: DECORUM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Samuel Demaria Jr, Professor, Anesthesiology Perioperative and Pain Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY-21-00270
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Postpartum Recovery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conversation (Experimental): Scripted interaction
  Interventions: Other: Disparities Conversation
- No Conversation (No Intervention): Control Group

INTERVENTIONS:
Other: Disparities Conversation — The study intervention will be a scripted interaction delivered by an anesthesia healthcare provider to an individual patient admitted to the labor/delivery unit for labor epidural placement and obstetric care. The discussion will highlight current data relating to healthcare disparities in obstetric anesthesia care within underserved groups and will explain various aspects of obstetric anesthesia care in a culturally-sensitive manner.
  Arms: Conversation

SUMMARY:
Racial and ethnic disparities in obstetric anesthesia care remains persistent despite studies documenting its existence and calling for action. The goal of this study is to share disparity data with underserved minority groups being admitted to the labor and delivery unit for obstetric care, to reduce mistrust and misconceptions regarding obstetric anesthesia care, and to bridge the cultural gap between patient beliefs and safe anesthetic care and to empower patients through transparency and provide them with the information necessary to make informed decisions about their care, to improve health literacy, and to ultimately improve patient outcomes and satisfaction.

DETAILED DESCRIPTION:
Patients admitted to Labor and Delivery Unit at MSH will self-identify race/ethnicity as part of the standard admission process (Documented in EPIC). Patients who elect for epidural placement for labor epidural analgesia will be approached by an Anesthesia Team Member to be enrolled in a minimal risk study. Participants who self-identify as a racial/ethnic underserved group (as defined by the NIH) will be randomized to receive routine care with a disparities discussion or routine care alone (in a Block Randomization format). Self-identified white participants will receive routine care and serve as a secondary comparison group. The disparities discussion will be performed following epidural placement when the patient is comfortable. During the postpartum period at patient follow-up (within 24hrs postpartum), an 18-point questionnaire evaluating outcomes and patient satisfaction will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Parturient patients being admitted to the labor and delivery unit at The Mount Sinai Hospital.
* Patients of age 18 or greater with a singleton fetus of at least 37 weeks of gestation that present in spontaneous labor, for induction of labor, or augmentation of labor.
* Patients in the first stage of labor and who have consented for placement of a labor epidural.

Exclusion Criteria:

* Patients who are in severe labor pain following verbal informed consent prohibiting them from participating in the discussion,
* Patients who present with a coagulopathy or on anticoagulation medications that exclude them from receiving labor epidural analgesia,
* Patients who do not consent to labor epidural placement, or if they are on a mid-wife service.
* Patients that are converted to a cesarean delivery following trial of labor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
DECORUM Questionnaire | postpartum Day 1
  DECORUM Questionnaire is split into 2 subscales, scored separately: The first subscale are built from the Obstetric-Quality of Recovery-10 Questionnaire scored from 0-100, with higher score indicating better health outcomes. The second subscale built from the Maryland Cultural Competency Questionnaire scored from 8 - 80, with higher score indicating better health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel DeMaria Jr., MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Allen Ninh, MD, Study Director — Icahn School of Medicine at Mount Sinai; Daniel Katz, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- The Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.